CLINICAL TRIAL: NCT03584698
Title: The Effect of Adding Vaginal Evening Primrose Oil to Misoprostol During Induction of Second-trimester Missed Miscarriage; a Randomized Controlled Trial
Brief Title: Evening Primrose Oil to Misoprostol During Induction of Second-trimester Missed Miscarriage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPOM
Record Dates: First submitted 2018-06-30; First posted 2018-07-12 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed | interventions — Misoprostol; evening primrose oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Misoprostol + Evening primrose oil group
  Interventions: Drug: Misoprostol 100Mcg Tab; Drug: Evening Primrose Oil 1000 MG
- control group (Active Comparator): Misoprostol only group
  Interventions: Drug: Misoprostol 100Mcg Tab

INTERVENTIONS:
Drug: Misoprostol 100Mcg Tab — women will receive misoprostol 100 mcg (Misotac, Sigma Pharmaceuticals, Egypt) vaginally applied every 6 hours till cervical dilatation.
Drug: Evening Primrose Oil 1000 MG — women will receive 4 capsules evening primrose oil 1000 mg (Primrose plus, Ema Pharm, Egypt) vaginally applied every 6 hours till cervical dilatation.
  Arms: study group

SUMMARY:
Termination of pregnancy is an important subject that has complex and emotional controversies. The most common time of termination of pregnancy is the mid-trimester which has two-thirds of all serious abortion-related complications. There are many indications for mid trimester termination of pregnancy such as missed abortion, serious fetal abnormalities and lastly some women do not wish to continue a pregnancy and will often request termination of pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Nullipara or previous vaginal delivery only
* Bishop score was ≤ 5
* Women who will accept to participate in the study

Exclusion Criteria:

* Multiple gestations
* Rupture of fetal membranes
* Previous cesarean sections
* Women with heavy bleeding
* Evidence of low implanted placenta by US
* Evidence of intra-uterine infection (either clinical or laboratory)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The induction to fetal expulsion time. | 24 hours
  Duration of delivery of fetus

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt